CLINICAL TRIAL: NCT04108182
Title: A Registry Study of Biomarkers in Progression of Acute Heart Failure
Brief Title: A Registry Study of Biomarkers in Progression of Acute Heart Failure(BIOMS-POAHF)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMS-POAHF
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Diseases
Keywords: heart failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The registry study aims to discover the prognostic value of bio-markers in acute heart failure

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged greater than or equal to 18 years with acute exacerbation of chronic heart failure or new heart failure
* 2. With typical symptoms of acute heart failure as follows: Dyspnea, ankle swelling and fatigue (Limited activity endurance), increased jugular pressure, rales and peripheral edema ;
* 3. Plasma concentrations of BNP: BNP>100pg/ML
* 4. Echocardiography: Related structural heart disease (left ventricular hypertrophy and/or left atrial enlargement) and/or diastolic dysfunction

Exclusion Criteria:

* 1. Previous history of cancer or renal replacement therapy
* 2.Surgery was performed within a month
* 3.Accompanied by cardiogenic shock, sepsis, pneumonia
* 4.Eligible patients without informed consent form

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure accorrding to Inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of death ( all cause) or readmission for heart failure | a median follow-up of 8.8 months
  Number of Death or heart failure related hospitalization within a median follow-up of 8.8 months of discharge

SECONDARY OUTCOMES:
Number of death ( all cause) or readmission for heart failure and cardiovascular mortality | a median follow-up of 8.8 months
  Number of Death or heart failure related hospitalization and cardiovascular mortality within a median follow-up of 8.8 months of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, PHD, Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

REFERENCES:
- [Derived] Ma K, Yang J, Shao Y, Li P, Guo H, Wu J, Zhu Y, Zhang H, Zhang X, Du J, Li Y. Therapeutic and Prognostic Significance of Arachidonic Acid in Heart Failure. Circ Res. 2022 Apr;130(7):1056-1071. doi: 10.1161/CIRCRESAHA.121.320548. Epub 2022 Mar 8. PMID 35255710